CLINICAL TRIAL: NCT04222790
Title: A Multicenter, Double-blind, Randomized Controlled Phase II Clinical Study of Monosialic Gangliosides to Prevent Albumin-bound Paclitaxel Neurotoxicity
Brief Title: A Study of Monosialic Gangliosides to Prevent Albumin-bound Paclitaxel Neurotoxicity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Zhenzhen Liu, Director, Henan Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HELEN-004
Record Dates: First submitted 2020-01-07; First posted 2020-01-10 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Early Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- monosialic ganglioside (Experimental): On the days -1, 1, and 2 of albumin paclitaxel application, 80 mg of monosialic ganglioside were applied (monosialic ganglioside was a single infusion)
  Interventions: Drug: monosialic gangliosides
- Placebo (Placebo Comparator): The control group received placebo on days -1, 1, and 2 of albumin paclitaxel (placebo as a single infusion)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: monosialic gangliosides — The experimental group received 80 mg of monosialic gangliosides (GM1) on days -1, 1, and 2 of albumin paclitaxel (GM1 is a single infusion).
  Other Names: experience group
  Arms: monosialic ganglioside
Other: Placebo — The control group received placebo on days -1, 1, and 2 of albumin paclitaxel (placebo as a single infusion)
  Other Names: control group
  Arms: Placebo

SUMMARY:
Taxane-induced peripheral neuropathy (TIPN) caused by paclitaxel is a dose-limiting toxicity. The main symptoms of discomfort are numbness, tingling, and burning sensations in the glove-sock-like distribution of the limbs. At present, there are few effective methods for clinical treatment of TIPN, and there is no widely agreed consensus on effective treatment in the world. Therefore, it is of great clinical significance and practical value to carry out clinical research to explore drugs to relieve TIPN.

DETAILED DESCRIPTION:
Taxane induced peripheral neuropathy (TIPN) caused by taxol is a dose limiting toxicity. The discomfort symptoms mainly include numbness, tingling and burning sensation in the glove sock like distribution of the extremities. This symptom can lead to limited activity, damage the self-care ability and social function of patients, and significantly reduce the quality of life of patients, At the same time, it may lead to early termination of chemotherapy and affect tumor treatment. The overall incidence of TIPN is very high. Many studies show that the incidence of TIPN is as high as 80%. CTCAE classifies it into 5 grades, and 25% - 30% of patients can have serious neurotoxicity. However, there are few effective methods for clinical treatment of TIPN, and there is no international consensus on effective treatment. Therefore, it is of great clinical significance and practical value to carry out clinical research on drugs to alleviate TIPN.

Monosialoganglioside (GM1), a member of the ganglioside family, is a kind of glycosylsphingolipid containing sialic acid on the cell membrane of mammalian animals. It is an endogenous substance. Gangliosides are mainly distributed in the outer layer of the cell membrane, especially on nerve endings and dendrites. It is most abundant and mainly expressed in the cell membrane of neurons. It participates in a variety of neurobiological activities, including neuronal differentiation Plasticity and cell survival. There is evidence that the application of GM1 can protect nerve cells, promote the recovery of neural function, and reduce the time of disability. Recent clinical studies on gangliosides have also shown promising results. GM1 effectively alleviates the neurotoxicity caused by docetaxel.

Although there have been previous studies on the effect of gangliosides on relieving the neurotoxicity of docetaxel, studies on the effect of gangliosides on relieving albumin bound paclitaxel have not been seen, and prospective clinical research data of large samples are lacking. In conclusion, the researchers hope to explore effective and reliable drugs to alleviate the peripheral neurotoxicity of albumin bound paclitaxel.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients diagnosed with early breast cancer by histology;
2. Age ≥18 years old and ≤75 years old
3. It is expected that the standard chemotherapy regimen containing albumin paclitaxel will be used in the adjuvant / neo-adjuvant chemotherapy regimen. The standard scheme includes: a. Albumin paclitaxel adopts a single-week regimen, 125-150mg / m2 for 12 weeks; b. Albumin paclitaxel Take a 3-week regimen, 260 mg / m2, for a total of 4 cycles. The plan must not contain platinum and other types of purple shirt drugs;
4. ECOG score of the patient is ≤1;
5. Expected survival time ≥ 3 months;
6. The function level of main organs must meet the following requirements (no blood transfusion and no use of leukocyte or platelet rising drugs within 2 weeks before screening) Blood routine: neutrophil (ANC) ≥ 1.5x 109 / L; platelet (PLT) ≥ 90x109 / L; hemoglobin (Hb) ≥ 90g / L Blood biochemical total bilirubin (TBIL) ≤ 1.5xULN; alanine aminotransferase (AST) and aspartate aminotransferase (AST) not exceeding 2 × ULN; blood urea nitrogen (BUN) and creatinine (CR) below 1.5 × ULN;
7. FACT-Ntx score is 44 points in the screening period
8. Sign the informed consent.

Exclusion Criteria:

1. There are any toxic events of the peripheral nervous system before enrollment, including: FACT-Ntx subscale score <44; ≥ 1 level of peripheral toxicity according to the CTCAE version 4.0 scale; all other pathological symptoms or diseases may affect Assessment of adverse neurotoxic effects;
2. Patients receiving other medications may cause similar adverse neurotoxic effects within 4 weeks before treatment with this regimen, or they may also receive neurotoxic medications at the same time. Including paclitaxel or analogues; vinca alkaloids or analogues; platinums or analogues; cytarabine, thalidomide, bortezomib or cabazine; other drugs or treatments may cause peripheral neurotoxicity;
3. Patients with poor overall condition and ECOG score> 1;
4. pregnant or lactating women;
5. Patients who also suffer from other neurological abnormalities cannot accurately record the occurrence and severity of neurotoxicity;
6. The patient is known to be allergic to the test drug or excipient ingredients of these products;
7. Patients with hereditary abnormalities of glucose and lipid metabolism (gangliopathies, such as idiopathic and retinopathy of triad families);
8. Patients not suitable for ganglioside treatment;
9. Patients with severe concurrent diseases may endanger safety and interfere with scheduled treatment, or the combination of diseases may affect the completion of the study, depending on the judgment of the investigator.
10. Patients with a clear history of neurological or mental disorders, including epilepsy or dementia.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2022-04-21 (Actual); Study Completion 2022-04-21 (Actual)

PRIMARY OUTCOMES:
Functional Assessment of Cancer Treatment Neurotoxicity Scale （FACT-Ntx）score | 2 weeks after 4 cycles of albumin-bound paclitaxel chemotherapy
  FACT-Ntx scale score 2 weeks after 4 cycles of albumin-bound paclitaxel chemotherapy. (The FACT-Ntx subscale includes 11 items, each of which is divided into 5 scoring levels: 0, 1, 2, 3, 4, and a total score of 44. Higher scores indicate lower side effects). The scale is graded 0-4. A low score indicates a good effect.

SECONDARY OUTCOMES:
CTCAE Version 4.0 score | 1 month Day 1 of Week 1 to 1 year after the last course of chemotherapy
  neurotoxicity evaluated by NCI-CTCAE version 4.0 grading scale which classified symptoms as grade 0, 1, 2, 3, or 4. Higher scores indicate more severe neurotoxicity.
  The NCI-CTCAE version 4.0 assessments were performed at 2 weeks after each course of chemotherapy. Additional long-term assessments were performed at 3 months, 6 months and 1 year after the end of chemotherapy.
Functional Assessment of Cancer Treatment Neurotoxicity Scale （FACT-Ntx）score | 3 months, 6 months, and 12 months after 4 cycles of chemotherapy
  The scale is graded 0-4. A low score indicates a good effect.
functional assesment of cancer therapy-taxane （FACT-Taxane）score | 2 weeks after 4 cycles of albumin-bound paclitaxel chemotherapy
  Compare FACT-Taxane outcome in treatment vs placebo groups at 2 weeks after 4 cycles of chemotherapy. Lower scores indicate worse functional status. Total possible range is 0 to 64.The paclitaxel therapeutic function assessment scale is mainly used to assess baseline peripheral neurotoxicity, and a lower score indicates less neurotoxicity.
Functional Assessment of Cancer Therapy-General （FACT-G）score | 2 weeks after 4 cycles of albumin-bound paclitaxel chemotherapy
  Compare FACT-G outcome in treatment vs placebo groups at 2 weeks after 4 cycles of chemotherapy. Lower scores indicate worse functional status. Total possible range is 0 to 128.The low score of the cancer patients' quality of life scale indicates that the patients' quality of life is better.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenzhen Liu, Study Director — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China